CLINICAL TRIAL: NCT00482885
Title: The Effect of Position on Oesophageal Peristalsis and LOS Pressures: a High Resolution Manometry Study
Brief Title: Coordination Versus Pressure in Oesophageal Peristalsis
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Dr Rami Sweis, St Thomas' Hospital
Other Study IDs: 07/Q0702/3
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Gastroesophageal Reflux
Keywords: Esophagus; Peristalsis; Contractile Pressure; Coordination of contraction; Bolus transport; Esophageal function
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
High Resolution Manometry (HRM) is a new advance in oesophageal measurement that permits the acquisition of pressure data through the entire length of the oesophagus over time via closely spaced sensors that continuously record the motor activity of the oesophagus. This allows not only contractile pressure to be measured, but also the coordination (proximal-distal) of contractions and the development of effective intra-bolus pressure (the force that drives bolus movement).

The study hypothesis is that (1) there will be a progressive increase in peristaltic pressure and decrease in velocity as the subjects move from the upright, through the supine to the upside down position and (2) the increase in pressure will be most evident in the mid-oesophagus at the transition zone between the striated and the smooth muscle contractions.

DETAILED DESCRIPTION:
Introduction High Resolution Manometry (HRM) is an advance in oesophageal measurement that permits the acquisition of pressure data through the entire length of the oesophagus over time via closely spaced sensors that continuously record the motor activity of the oesophagus. This information can then be analysed either as conventional line plots or as a spatiotemporal plot, a compact, visually intuitive presentation of oesophageal pressure activity.1 This process has been quantified and verified in 75 normal volunteers.2 Increasing evidence suggests that HRM is a more sensitive and accurate means of assessing oesophageal function compared to conventional manometry.1 3 Compared to conventional manometry, HRM increases the accuracy with which the success of bolus transport can be predicted.1 This is important because oesophageal symptoms are more closely linked to impaired bolus transport than conventional pressure measurements per se.4

The additional information provided by HRM and the presentation of data as a spatiotemporal plot enable investigators to study the pressure activity in the oesophagus during normal eating behaviour for the first time. This study will assess the effects of position, bolus volume and consistency (liquid, solid). In addition, pressure activity during a standardized test meal will be observed.

Understanding the oesophageal response due to these 'physiologic challenges' is likely to be of clinical importance because most patients complain of swallowing problems, regurgitation or chest pain during such events and in the postprandial period. This is in contrast to standard manometry protocols that include the intake only of individual water, viscous fluid (e.g. yoghurt) or small, solid bolus swallows.

Healthy controls will be studies to provide normal data. Patients referred for investigation of oesophageal symptoms will be studied to assess whether physiologic challenge increases the ability to differentiate this group from normal controls, explain patient symptoms and increase diagnostic yield.

Effects of Position It is well known that transient lower oesophageal sphincter relaxations (TLOSRs) and reflux events are suppressed in the supine position in both healthy volunteers and in patients with mild-moderate reflux disease.7 The effects of position on oesophageal peristalsis and lower oesophageal sphincter pressure assessed by conventional manometry have been less consistent.

Recently HRM and video-fluoroscopy has been applied to study the effect of position and bolus consistency on oesophageal function.8 No effect of position on LOS pressure was found in these thin, healthy volunteers. In contrast peristaltic pressure increased and velocity decreased as the subject moved from the upright to the supine position. Similarly, peristaltic pressure increased and velocity decreased progressively as the subject took dry, water and solid swallows.8 These observations confirm combined manometry and impedance studies that show oesophageal function is not stereotyped but responds to the workload required for bolus transport. 5 67

Although findings are consistent for a given individual, variation in peristaltic contractile pressure is high and the correlation between peristaltic pressure and the success of bolus transport in healthy volunteers and patients is weak. Rather, preliminary observations by Fox et al. suggest that successful bolus transport, especially for solids, may depend more on effective coordination between proximal (striated) and mid-distal (smooth muscle) contractions than increased peristaltic pressure. In particular the prompt response of the mid-oesophageal segment appears to be linked to successful bolus transport through the oesophagus.8

Swallowed material can be transported successfully through the oesophagus in the upside down position. With the use of HRM, a detailed analysis of oesophageal peristalsis and bolus transport from the pharynx to the stomach is possible. We propose to explore the effect of 3 different positions (upright, supine and 60o head down) on the swallow of liquid and viscous material in healthy volunteers. Use of the extreme head down position provides a classical physiologic challenge that will highlight the oesophageal response to increased work against gravity.

Further events that increase oesophageal workload include the rapid intake of large volumes of fluid (i.e. free drinking) and the intake of solid food (i.e. test meal). Following the studies of position on oesophageal function, we will then assess the effect of drinking a standardized fluid load by multiple repeated swallows and intake of a standardized test meal on oesophageal and lower oesophageal sphincter function. Observations will be continued for 20minutes after ingestion to assess also oesophago-gastric function in the postprandial period.

Study hypothesis The driving force developed by oesophageal motor function 'increases' progressively with workload (e.g. increasing inclination, solid food) in healthy volunteers.

Hypothesis #1: This 'increase in driving force' will be more apparent and consistent as an increased in coordination of peristaltic contractions and development of intra-bolus pressure (i.e. endpoints assessed only by HRM) than effects on contractile pressure (i.e.; endpoints assessed also by conventional manometry).

Repeated swallowing during drinking suppresses oesophageal contractility. Hypothesis #2: Intermittent, coordinated and powerful peristaltic waves will be observed during a test meal and failure of this activity will result in raised intra-bolus pressure and symptoms (dysphagia, regurgitation, chest pain).

Hypothesis #3: Observations during and after a test meal will increase diagnostic yield for rumination and reflux related symptoms during stationary studies.

ELIGIBILITY:
Inclusion criteria

Subjects to be included in the study are those:

1. male or female
2. at least 18 years of age
3. have given informed consent for the HRM procedure

Exclusion Criteria

For normal controls:

1. with symptoms or a history of oesophageal gastrointestinal disease
2. with regular intake of medication. Occasional use of analgesic (e.g. aspirin) is allowed
3. with any hematological abnormalities
4. with any evidence of infectious disease
5. who are pregnant or breast-feeding.
6. with evidence or history of drug or alcohol abuse within the past two years
7. with diabetes mellitis
8. with mental impairment limiting the ability to comply with study requirements
9. who are taking or planning to take other investigational drugs during the study
10. with use of medications influencing upper GI motility within one week of the study (i.e. calcium channel blockers, prokinetic drugs, macrolide antibiotics).
11. with use of PPIs and H2 blockers

For patients:

1. with no oesophageal symptoms (e.g. referred for studies prior to bariatric surgery)
2. with mental impairment limiting the ability to comply with study requirements
3. who are taking or planning to take other investigational drugs during the study
4. with use of medications influencing upper GI motility within one week of the study (i.e. calcium channel blockers, prokinetic drugs, macrolide antibiotics).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and patients presenting with symptoms of reflux and endoscopy negative dysphagia
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fox, MD, Principal Investigator — Honorary Consultant and Senior Lecturer
Locations (1):
- Oesophageal Laboratory, GSTT, London, London, United Kingdom